CLINICAL TRIAL: NCT04947215
Title: The Association Between LPCAT1 Genetic Polymorphism and Stress Biomarkers in Neonatal Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Elrasoul Sayed, clinical pharmacist, Assiut University
Other Study IDs: Neonatal RDS
Record Dates: First submitted 2021-06-14; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Neonatal Respiratory Distress
Keywords: LPCAT 1
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Two and half mL of cord blood will be obtained from umbilical cord artery immediately after delivery on tube after centrifugation the serum will be separated and frozen at -70oC until analysis of stress biomarker.
  * Two and half mL of peripheral blood will be obtained from neonates on EDTA tube that was preserved at -70 C for DNA extraction for genetics work.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases group: It includes 100 neonates who are admitted in the neonatal intensive care unit in Assiut University children hospital suffering from RDS. The cases will be subdivided into subgroups according to1. Full term or preterm, 2. Type of pregnancy (normal or complicated), 3. Mode of delivery, and 4. LPCAT1 genetic polymorphism.
  Interventions: Diagnostic Test: stress biomarkers
- control group: include 60 neonates without RDS.
  Interventions: Diagnostic Test: stress biomarkers

INTERVENTIONS:
Diagnostic Test: stress biomarkers — used to estimate the reference values of putative biomarkers of birth stress such asCTnT, CTnI, copeptin, NT-proBNP and hs-CRP in the cord blood of full term neonates

SUMMARY:
Aims of the Research

Primary:

1. Measure the levels of stress biomarkers in full and preterm neonates with normal and complicated pregnancies and to study the influence of delivery mode on their cord blood concentrations.
2. Test the association between LPCAT1 genetic polymorphism and the levels of these biomarkers in neonates suffering from RDS.
3. Study the relation between LPCAT1 genetic polymorphism and the risk/severity of neonatal respiratory distress syndrome.

Secondary:

1) Help understanding the possible etiology and pathogenesis of neonatal RDS. 2) Help the possibility of early detection, diagnosis and management.

3) Help to decrease mortality and morbidity in selective cases. 4) Understand the individual variability in the susceptibility to development of pulmonary pathologies.

DETAILED DESCRIPTION:
Neonatal respiratory distress syndrome (RDS) is caused by lung immaturity and deficiency of lung surfactant and dysfunction in preterm newborns . Surfactant is produced by type II pneumocyte that forms a bilayer of lipid over the inner surface of the alveoli. Surfactant deficiency and dysfunction lead to increased alveolar surface tension, which results in alveolar collapse and decreased lung aeration . Respiratory distress syndrome is one of the main causes of neonatal mortality . The risk of RDS increases with decreasing gestational age (GA). The incidence of RDS was estimated to be 90% in preterm neonates (GA 28 weeks or below) and to be 9% in full term neonates born at ≥38 weeks' gestation. Early diagnosis is very essential to optimize the treatment of infants with RDS.

Pathogenesis The primary cause of RDS is deficiency and/or dysfunction of surfactant which is a lipoprotein complex and is vital for normal lung function. Surfactant is synthesized, stored, and secreted by the alveolar type II cells and is primarily composed of phospholipids, which constitute 80-85% of the total mass. The remaining components of surfactant includes neutral lipids (5%-10%) and proteins (10%) . Phosphatidylcholine (PC), the most abundant phospholipid species in surfactant, constitutes 80% of the total phospholipids. There are three key enzymes involved in the PC synthesis: Lysophospholipid acyltransferase (LPCAT1, Gene ID 79888), Cholinephosphotransferase (CHPT1, Gene ID 56994) and Cholinephosphate cytidylyltransferase (PCYT1B, CPCT, Gene ID 9468). LPCAT1 is the most important enzyme in biogenesis and a key enzyme in surfactant production . LPCAT1 composed of 18 exons and is located on chromosome 5p15.33. The study of the genetic polymorphisms of surfactant-lipids related gene provides significant data about individual variability in the susceptibility to development of respiratory distress syndrome.

Neonatal stress biomarkers such as cardiac troponin (CTn) T, CTnI, NT-Terminal-pro-Brain Natriuretic Peptide (NT-pro-BNP), copeptin, and high sensitivity C-reactive protein (hs-CRP)have been considered as an indicator of perinatal asphyxia. Troponin is an inhibitory protein complex located on the actin filament in all striated muscle and consists of three subunits: T, C, and I. The asphyxiated neonate has elevated levels of cardiac troponin I (cTnI). cTnI is thought to be also an indicator of perinatal asphyxia . Neonates born after complicated delivery had significantly higher values of CTnT, CTnI and Copeptin than those born after uncomplicated delivery. The gender influence on copeptin releases . The gestational age, birth weight and duration of active labor, and membrane rupture have significant effect on hs-CRP levels.

ELIGIBILITY:
Inclusion Criteria:

* neonates who are admitted in the neonatal intensive care unit in Assiut University children hospital suffering from RDS.

Exclusion Criteria:

* The newborn will be excluded from the study when his/her parents refuses to participate or when the neonate presented with one or more of the following:

  1. Multiple congenital anomalies
  2. Severe infection
  3. Inherited metabolic disorders
  4. Any systemic disorder (hepatic, renal, cardiovascular, and endocrinal, ...etc)
  5. Malignancies
  6. Hypoxic Ischemic Encephalopathy

Ages: 1 Hour to 1 Month | Sex: All
Age Groups: Child
Study Population: A case-control study
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
LPCAT1 genetic polymorphism | "1 year"
  The LPCAT1genetic polymorphism work will be performed using an improved multiplex ligation detection reaction (iMLDR) technique .Genomic DNA from patients will be extracted from peripheral blood by DNA mini extraction kit.

SECONDARY OUTCOMES:
The electrochemiluminescence immunoassay ECLIA: | "1 month"
  This method will be used to estimate the reference values of putative biomarkers of birth stress CTnT in the cord blood of full term neonates
The electrochemiluminescence immunoassay ECLIA | "2 month"
  This method will be used to estimate the reference values of putative biomarkers of birth stress hs-CRP in the cord blood of full term neonates

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut university, Asyut
  - Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bisschop B, Derriks F, Cools F. Early Predictors for INtubation-SURfactant-Extubation Failure in Preterm Infants with Neonatal Respiratory Distress Syndrome: A Systematic Review. Neonatology. 2020;117(1):33-45. doi: 10.1159/000501654. Epub 2019 Aug 22. PMID 31437836
- [Background] Ma H, Yan W, Liu J. Diagnostic value of lung ultrasound for neonatal respiratory distress syndrome: a meta-analysis and systematic review. Med Ultrason. 2020 Sep 5;22(3):325-333. doi: 10.11152/mu-2485. Epub 2020 Apr 15. PMID 32399541
- [Background] Alemu AY, Belay GM, Berhanu M, Minuye B. Determinants of neonatal mortality at neonatal intensive care unit in Northeast Ethiopia: unmatched case-control study. Trop Med Health. 2020 Jun 3;48:40. doi: 10.1186/s41182-020-00232-9. eCollection 2020. PMID 32514229
- [Background] Kim M, Porras-Gomez M, Leal C. Graphene-based sensing of oxygen transport through pulmonary membranes. Nat Commun. 2020 Feb 27;11(1):1103. doi: 10.1038/s41467-020-14825-9. PMID 32107376
- [Background] Lin S, Ikegami M, Moon C, Naren AP, Shannon JM. Lysophosphatidylcholine Acyltransferase 1 (LPCAT1) Specifically Interacts with Phospholipid Transfer Protein StarD10 to Facilitate Surfactant Phospholipid Trafficking in Alveolar Type II Cells. J Biol Chem. 2015 Jul 24;290(30):18559-74. doi: 10.1074/jbc.M115.666701. Epub 2015 Jun 5. PMID 26048993
- [Background] Shen W, Kuang P, Wang B, Zeng Q, Chen C, Lin X. Genetic Polymorphisms of LPCAT1, CHPT1 and PCYT1B and Risk of Neonatal Respiratory Distress Syndrome among a Chinese Han Population. Pediatr Neonatol. 2020 Jun;61(3):318-324. doi: 10.1016/j.pedneo.2019.12.012. Epub 2020 Jan 3. PMID 31964590
- [Background] Rouatbi H, Zigabe S, Gkiougki E, Vranken L, Van Linthout C, Seghaye MC. Biomarkers of neonatal stress assessment: A prospective study. Early Hum Dev. 2019 Oct;137:104826. doi: 10.1016/j.earlhumdev.2019.104826. Epub 2019 Jul 27. PMID 31362253
- [Background] Evers KS, Wellmann S. Arginine Vasopressin and Copeptin in Perinatology. Front Pediatr. 2016 Aug 2;4:75. doi: 10.3389/fped.2016.00075. eCollection 2016. PMID 27532032
- [Background] Ishibashi M, Takemura Y, Ishida H, Watanabe K, Kawai T. C-reactive protein kinetics in newborns: application of a high-sensitivity analytic method in its determination. Clin Chem. 2002 Jul;48(7):1103-6. No abstract available. PMID 12089183